CLINICAL TRIAL: NCT01931163
Title: Neoadjuvant Phase II Study Of Everolimus Plus Cisplatin In Triple Negative Breast Cancer Patients With Residual Disease After Standard Chemotherapy
Brief Title: NECTAR Everolimus Plus Cisplatin in Triple (-) Breast Cancer
Acronym: NECTAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jenny C. Chang, MD (Other)
Collaborators: The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor-Investigator, Jenny C. Chang, MD, Sponsor-Investigator/Principal Investigator, The Methodist Hospital Research Institute
Organization: The Methodist Hospital Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00008952; IRB(2)#0513-0062 (Other: TMHRI IRB); CRAD001 JUST213 (Other: Other ID)
Record Dates: First submitted 2013-08-26; First posted 2013-08-29 (Estimated); Results first posted 2021-07-09 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Breast Cancer; Triple Negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Everolimus (Experimental): Cisplatin 20 mg/m2 IV infusion over 60 minutes, weekly (Days 1, 8, 15) x 4 cycles Everolimus 10mg by mouth daily
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus
  Other Names: RAD001; Afinitor

SUMMARY:
RATIONALE: Everolimus plus Cisplatin may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: The purpose of this study is to test how effective combining Cisplatin chemotherapy with Everolimus is in treating subjects with triple negative breast cancer who have residual disease after chemotherapy.

DETAILED DESCRIPTION:
This is a phase II clinical trial of everolimus, an mTOR inhibitor, plus cisplatin chemotherapy in patients with triple negative breast cancer (TNBC) who have residual disease after completion of neoadjuvant chemotherapy. Everolimus and cisplatin will be administered for 12 weeks. Patients will undergo surgery after treatment completion. Patients will have breast biopsy prior to receiving the study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients ≥18 years of age.
2. Clinical/pathological documentation of residual disease after neo-adjuvant therapy.
3. Patients with synchronous bilateral cancers are eligible only if:

   • Index cancer is triple-negative, defined as ER-, PR-, and HER2-.
4. HER2 negative tumors. HER2 negativity must be confirmed by one of the following:

   * FISH-negative (FISH ratio <2.2), or
   * IHC 0-1+, or
   * IHC 2-3+ AND FISH-negative (FISH ratio <2.2).
5. Estrogen receptor negative and progesterone receptor negative (<10% staining by IHC for estrogen receptor and progesterone receptor).
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
7. Adequate hematologic function, defined by:

   * Absolute neutrophil count 2 >1000/mm3
   * Platelet count ≥100,000/mm3
   * Hemoglobin >9 g/dL
8. Adequate liver function, defined by:

   * AST and ALT ≤2.5 x the upper limit of normal (ULN)
   * Total bilirubin ≤1.5 x ULN (unless the patient has grade 1 bilirubin elevation due to Gilbert's disease or a similar syndrome involving slow conjugation of bilirubin).
9. Adequate renal function, defined by:

   • Serum creatinine ≤1.5 x ULN
10. Complete staging work-up ≤24 weeks prior to initiation of study treatment with computed tomography (CT) scans of the chest and abdomen/pelvis (abdomen/pelvis preferred; abdomen accepted), a CT scan of the head or MRI of the brain (if symptomatic), and either a positron emission tomography (PET) scan or a bone scan.
11. Adequate cardiac function, defined by a left ventricular ejection fraction (LVEF) value of >50% (or normal per institutional guidelines) by MUGA scan or echocardiogram (ECHO).
12. Patients with previous history of invasive cancers (including breast cancer) are eligible if definitive treatment was completed more than 5 years prior to initiating current study treatment, and there is no evidence of recurrent disease.
13. Women of childbearing potential must have a negative serum or urine pregnancy test performed within 7 days prior to start of treatment. If a woman becomes pregnant or suspects she is pregnant while participating in this study, she must agree to inform her treating physician immediately.
14. Patient must be accessible for treatment and follow-up.
15. Women of childbearing potential must agree to use an acceptable method of birth control to avoid pregnancy for the duration of study treatment, and for 3 months thereafter.
16. Able to swallow and retain oral medication.
17. Patient must be willing to undergo breast biopsies as required by the study protocol.
18. All patients must be able to understand the investigational nature of the study and give written informed consent prior to study entry.

Exclusion Criteria:

1. Women who are pregnant or breastfeeding.
2. History of previously treated ductal carcinoma in situ (DCIS) is acceptable.
3. Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel.
4. Known intolerance or hypersensitivity to Everolimus or other rapamycin analogs (e.g. sirolimus, temsirolimus);
5. Previous cancer (with the exception of non-melanoma skin cancer or cervical carcinoma in situ) in the past 5 years.
6. Patients who have any severe and/or uncontrolled medical conditions such as:

   1. unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction ≤6 months prior to start of Everolimus, serious uncontrolled cardiac arrhythmia, or any other clinically significant cardiac disease
   2. Symptomatic congestive heart failure of New York heart Association Class III or IV
   3. active (acute or chronic) or uncontrolled severe infection, liver disease such as cirrhosis, decompensated liver disease, and chronic hepatitis (i.e. quantifiable HBV-DNA and/or positive HbsAg, quantifiable HCV-RNA),
   4. known severely impaired lung function (spirometry and DLCO 50% or less of normal and O2 saturation 88% or less at rest on room air),
   5. active, bleeding diathesis;
7. Patients may not receive any other investigational or anti-cancer treatments while participating in this study.
8. Concurrent severe, uncontrolled infection or intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements.
9. Mental condition that would prevent patient comprehension of the nature of, and risk associated with, the study.
10. Inability to comply with study and/or follow-up procedures.
11. Patients who have received live attenuated vaccines within 1 week of start of Everolimus and during the study. Patient should also avoid close contact with others who have received live attenuated vaccines.

    Examples of live attenuated vaccines include intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella and TY21a typhoid vaccines;
12. Known history of HIV seropositivity;
13. Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing of study treatment. Highly effective contraception methods include combination of any two of the following (a+b or a+c or b+c):

    1. Use of oral, injected or implanted hormonal methods of contraception or;
    2. Placement of an intrauterine device (IUD) or intrauterine system (IUS);
    3. Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/ vaginal suppository;
    4. Total abstinence or;
    5. Male/female sterilization. Women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks prior to treatment. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child-bearing potential.
14. Chronic treatment with corticosteroids or other immunosuppressive agents. Topical or inhaled corticosteroids are allowed;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-07; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Chang, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (3):
- United States (3):
  - The Methodist Hospital, Houston, Texas
  - Houston Methodist Hospital Willowbrook, Houston, Texas
  - Houston Methodist Hospital Sugar Land, Sugar Land, Texas

REFERENCES:
- [Derived] Anand K, Patel T, Niravath P, Rodriguez A, Darcourt J, Belcheva A, Boone T, Ensor J, Chang J. Targeting mTOR and DNA repair pathways in residual triple negative breast cancer post neoadjuvant chemotherapy. Sci Rep. 2021 Jan 8;11(1):82. doi: 10.1038/s41598-020-80081-y. PMID 33420229

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 24 patients with Stage II/III Triple Negative Breast Cancer with residual cancer >1cm post-neoadjuvant anthracycline and taxane-based chemotherapy were enrolled.
  Of the 24 patients, 2 were excluded (one because of metastasis before treatment and one because of withdrawal); 22 were included in the efficacy analysis.
Groups:
- Everolimus Plus Cisplatin: Cisplatin 20 mg/m2 IV infusion over 60 minutes, weekly (Days 1, 8, 15) x 4 cycles Everolimus 10mg by mouth daily
Period: Overall Study
Arm/Group | Everolimus Plus Cisplatin
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Everolimus Plus Cisplatin
Number analyzed (Participants) | 22
Age, Continuous [Median (Full Range); unit: years] | 50.1 [31.9 to 74.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 22
TNBC patients with residual cancer >1 cm post neoadjuvant anthracycline and chemotherapy [Count of Participants; unit: Participants] | 22

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response
Description: Evaluate tumor response using RECIST criteria after 12 weeks of treatment at definitive surgery.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.", or similar definition that is accurate and appropriate.
Time Frame: tumor response at 12 weeks after treatment
Measure: Count of Participants; unit: Participants
Groups:
- Everolimus Plus Cisplatin: Everolimus 10mg by mouth daily for 12 weeks; Cisplatin 20 mg/m2 IV infusion over 60 minutes, weekly (Days 1, 8, 15) x 4 cycles
Arm/Group | Everolimus Plus Cisplatin
Number analyzed (Participants) | 22
Participants | 22

ADVERSE EVENTS:
Time Frame: Data was collected during treatment period of 12 weeks
Arm/Group | Everolimus Plus Cisplatin
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 6/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus Plus Cisplatin (N=22)
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Nausea (General disorders) | 1
leucocytopenia (Blood and lymphatic system disorders) | 1
papilledema (Eye disorders) | 1
neutropenia (Blood and lymphatic system disorders) | 1
hyperglycemia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus Plus Cisplatin (N=22)
Nausea (General disorders) | 9
Fatigue (General disorders) | 10
Mucositis (General disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-04-28): https://cdn.clinicaltrials.gov/large-docs/63/NCT01931163/Prot_SAP_000.pdf